CLINICAL TRIAL: NCT00640952
Title: Acamprosate for Treatment of Compulsive Behaviors and Craving in Parkinson's Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left site
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Parkinson Foundation (Other)
Responsible Party: Principal Investigator, Joohi Jimenez-Shahed, Principal Investigator, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-19781
Record Dates: First submitted 2007-12-28; First posted 2008-03-21 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; impulse control behaviors; dopa-dysregulation
MeSH Terms: conditions — Parkinson Disease | interventions — Acamprosate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: acamprosate — 333 mg 2 tabs tid

SUMMARY:
The purpose of this study is to determine how many patients with Parkinson's disease have compulsive behaviors, and what types of behaviors they have. This study will also determine if acamprosate can be used to treat compulsive behaviors in Parkinson's disease patients.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic Parkinson's disease
2. Active dopaminergic therapy at stable dose for one month (levodopa or dopamine agonist)
3. Able and willing to complete Rating Scales
4. Presence of one or more compulsive behavior based on responses to Rating Scales (defined as >5 on the SOGS; >17 on the YBOCS-SV and YBOCS-CUV; >1.7 on the SCS for women and >2.1 on the SCS for men; >15 on the YBOCS-BE, >5.5 on the CQ).
5. Written informed consent

Inclusion criteria (controls):

1. No significant psychiatric disease
2. Able and willing to complete Rating Scales
3. Written informed consent

Exclusion Criteria:

1. No anticipated need for adjustment of medications for Parkinson's disease
2. Current participation in another clinical study
3. History of unstable psychiatric disease (as determined by the Principal Investigator)
4. Women of childbearing age not using appropriate contraceptive methods (oral contraceptives, condoms, surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
safety and efficacy compared to baseline scores | 6 months

SECONDARY OUTCOMES:
change from baseline assessment tools used in the study | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joohi Jimenez-Shahed, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- PDCMDC 6550 Fannin, Suite 1801, Houston, Texas, United States

REFERENCES:
- See also: Parkinson's Disease Center and Movement Disorders Clinic — http://www.jankovic.org